CLINICAL TRIAL: NCT01162226
Title: "PD Wii: Computer-based Gait and Balance Training for Parkinson's Patients".
Brief Title: Computer-Based Balance Training for People With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Glenna Dowling, RN, PhD, FAAN, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2R42NS061502-02 (NIH); 2R42NS061502-02 (NIH)
Record Dates: First submitted 2010-06-24; First posted 2010-07-14 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Parkinson's Disease
Keywords: gait; movement disorders; balance; function
MeSH Terms: conditions — Parkinson Disease; Movement Disorders | interventions — Gait

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- training program (Experimental)
  Interventions: Behavioral: gait and balance training program

INTERVENTIONS:
Behavioral: gait and balance training program — The intervention will be implemented via three 50-minute training sessions per week for 12 weeks. The games will be played when the subject is receiving the maximum benefit from their anti-parkinsonian medications. The control group and the intervention group will receive weekly telephone calls to inquire about medications and falls. At baseline and end of the 12 weeks, in-home testing will determine stride length and speed; standing balance eyes open and closed on flat and foam surface.

SUMMARY:
This study will be carried out to determine the effectiveness of in-home computer games played by a person with Parkinson's disease for 50 minutes 3 times a week on measures of standing and walking balance.

ELIGIBILITY:
Inclusion Criteria:

1. presence of bradykinesia along with at least one of the following: muscular rigidity, 4-6 Hz rest tremor, and postural instability (Gelb, Oliver, & Gilman, 1999; Hughes, Ben-Shlomo, Daniel, & Lees, 1992).
2. Hoehn & Yahr disease Stage 1 (unilateral disease) to 3 (mild to moderate bilateral disease, physically independent) (Fahn and Elton, 1987).

Exclusion Criteria:

1. history of strokes, repeated head injury, encephalitis, oculogyric crises, neuroleptic treatment, MPTP exposure, more than one affected relative, sustained remission, strictly unilateral features after 3 years, supranuclear gaze palsy, early severe autonomic involvement or dementia, Babinski sign, tumor, or a negative response to L-DOPA (Hughes et al., 1992).
2. other neurologic, orthopedic or cardiac problems, cognitive impairment as evidenced by 5 or more errors on the Mini Mental State Examination (MMSE) (Folstein, Folstein, & McHugh, 1975)
3. visual or hearing impairments serious enough to interfere with their ability to interact with the computer-based training program.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
gait | 3 months
  Gait velocity and stride length will be measured with WriteStep Gait and Mobility pads (Abilitations). For the gait analysis, subjects will walk along a 10 foot walkway (gait velocity) that will record the footprint patterns from which we will evaluate the time it takes to walk the distance of the walkway and the average stride length. Each subject will walk according to standard protocol of 1 trial at his/her self-selected speed to enable an accurate representation of usual gait.
balance | 3 months
  Balance will be objectively measured using the modified Clinical Test for Sensory Interaction and Balance (CTSIB) (Shumway-Cook & Horak, 1986). There are 2 conditions with a stable platform (eyes open and eyes closed) and 2 conditions on a less stable foam surface, (eyes open and eyes closed). Following the standardized protocol, subjects will be tested 3 times in each condition on the stable surface and 3 times in each unstable condition for up to thirty seconds each. The number of seconds standing will be summed across all 12 trials for a range of 0-360 seconds.

SECONDARY OUTCOMES:
falls | weeks 1-12
  Weekly phone inquiry will quantify number of falls if any, during the past week.
overall functional status | 3 months
  Functional status will be assessed by the Unified Parkinson's Disease Rating Scale (UPDRS, Parts 2 & 3) (Fahn, Elton, & Members of the UPDRS Committee, 1987). Part 2 is a quantitative 5-point scale that measures the subjects' perception of their functional status. Part 3 is also a 5-point scale in which a clinician evaluates actual functional status by physical exam. The scores on each item in Parts 2 & 3 are summed to yield a total score.
subjective balance | 3 months
  Subjective balance will be assessed by the Activities-specific Balance Confidence (ABC) Scale (Powell & Myers, 1995). This instrument assesses subjective balance/fear of falling by asking subjects to rate the degree of confidence that they have for completing 16 activities of daily living without falling. Ratings are summed and then divided by 16 (or the number of items completed) to yield a total ABC score.
balance | 3 months
  Timed up and go test (TUG) will be a secondary measure of balance. Subjects are seated in a straight back chair with arms. On the command "GO" the stop watch is started. Subject stands, walks toward a visible object on the floor positioned 8 feet from chair, walk around the object, return to chair and sit down. After a practice, 3 TUG will be performed. Times will be documented in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Glenna A Dowling, PhD, Principal Investigator — University of Ca San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Fahn, S., Elton, R., & Members, U. C. (1987). Unified Parkinson's disease rating scale. In S. Fahn, C. D. Mardsen, M. Goldstein & D. Calne (Eds.), Recent Developments in Parkinson's Disease (pp. 153-163). New Jersey: Macmillan Healthcare Information. Folstein, M. F., Folstein, S. E., & McHugh, P. R. (1975).
- [Background] Folstein MF, Folstein SE, McHugh PR.
- [Background] Gelb DJ, Oliver E, Gilman S. Diagnostic criteria for Parkinson disease. Arch Neurol. 1999 Jan;56(1):33-9. doi: 10.1001/archneur.56.1.33. PMID 9923759
- [Background] Hughes AJ, Ben-Shlomo Y, Daniel SE, Lees AJ. What features improve the accuracy of clinical diagnosis in Parkinson's disease: a clinicopathologic study. Neurology. 1992 Jun;42(6):1142-6. doi: 10.1212/wnl.42.6.1142. PMID 1603339
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Shumway-Cook A, Horak FB. Assessing the influence of sensory interaction of balance. Suggestion from the field. Phys Ther. 1986 Oct;66(10):1548-50. doi: 10.1093/ptj/66.10.1548. No abstract available. PMID 3763708